CLINICAL TRIAL: NCT00297011
Title: Valacyclovir+Temovate Gel for the Episodic Treatment of Herpes Labialis: A Patient-Initiated Double-Blind, Placebo-Controlled Study, Randomized Study.
Brief Title: Valacyclovir+Temovate Gel for the Treatment of Herpes Labialis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Christopher Hull, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 50301066
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Last update posted 2008-05-06 (Estimated); Status verified 2008-04

CONDITIONS: Herpes Labialis
MeSH Terms: conditions — Herpes Labialis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: valacyclovir+clobetasol gel

SUMMARY:
A randomized study comparing the combination of valacyclovir and temovate gel (clobetasol gel) versus placebo for the treatment of recurrent herpes labialis (cold sores).

DETAILED DESCRIPTION:
Herpes simplex labialis is a common, worldwide affliction for which neither public health procedures, vaccines, nor antiviral chemotherapy have had a major impact. The present study has been proposed because it has become clear there are marked limitations to the benefit of antiviral therapy in herpes labialis. Recently, a pilot trial of the combination of famciclovir and topical 0.05% fluocinonide vs famciclovir alone showed that the addition of corticosteroids to the antiviral drug treatment caused a marked and statistically significant reduction in lesion size and a trend to more aborted lesions.

This study is designed as a randomized, placebo-controlled, , patient-initiated study. The objective of this study is to evaluate the safety and efficacy of oral valacyclovir 2grams BID for one day and topical temovate 0.05% gel BID for three days compared to placebo capsules and placebo gel in the episodic treatment of a single episode of recurrent herpes labialis in immunologically normal patients.

Subjects will be screened, randomized to study drug and instructed to start using study drug within one hour of the first sign or symptom of their next episode of herpes labialis. Data on the treated lesion will be collected by clinic visits and a patient diary card.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* A history typical for recurrent herpes labialis. The subject must have experienced three or more cold sores in the last 12 months.
* In general good health, without other serious medical conditions, as determined by the patient's account of his/her medical history.
* Signature on the informed consent document.

Exclusion Criteria:

* Patients who have participated in an investigational drug study in the four-week period prior to enrollment.
* Previous herpes vaccine at any time.
* Patients with major medical conditions such as chronic heart, pulmonary, renal or hepatic diseases.
* Patients with immunodeficiency disorders such as HIV infection or cancer chemotherapy.
* Patients using topical steroids on or near the face or systemic steroids within 30 days of enrollment.
* Women who are pregnant, lactating or breast feeding.
* Women of childbearing potential not using adequate contraception as judged by the Investigator.
* Recent history of alcohol or drug abuse, which in the opinion of the investigator, may interfere with that study patient's compliance with study requirements.
* Significant skin disease such as atopic dermatitis, acne, or rosacea that would interfere with the assessment of lesions.
* Allergy or hypersensitivity to steroids, acyclovir, penciclovir and/or other nucleoside analogues.
* Subjects with impaired renal function as defined as a serum creatinine above the upper limits of normal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-09; Primary Completion 2007-03 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable is the maximum size of the primary lesion complex

SECONDARY OUTCOMES:
Secondary variables include: the proportion of primary lesions that are aborted; the mean time to healing of the primary lesion complex the frequency and mean duration of lesion pain among primary lesions; the frequency of secondary lesions

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hull, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Hull C, McKeough M, Sebastian K, Kriesel J, Spruance S. Valacyclovir and topical clobetasol gel for the episodic treatment of herpes labialis: a patient-initiated, double-blind, placebo-controlled pilot trial. J Eur Acad Dermatol Venereol. 2009 Mar;23(3):263-7. doi: 10.1111/j.1468-3083.2008.03047.x. Epub 2009 Jan 8. PMID 19143902